CLINICAL TRIAL: NCT05550519
Title: A Prospective Study to Investigate the Relationship Between Hepatitis B Surface Antigen (HBsAg) Loss and the Dynamics in Host and Viral Markers After Discontinuation of Nucleos(t)Ide Analog (NA) Treatment in Chronic Hepatitis B E-antigen Negative Patients With Low On-treatment HBsAg Level
Brief Title: A Study in Chronic Hepatitis B e-Antigen Negative Participants After Discontinuation of Nucleos(t)Ide Analog (NA) Treatment
Acronym: SALMONS
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision after re-evaluation of strategy in the context of recruitment timelines projection
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR109229; NOPRODHPB0017 (Other: Janssen Research & Development, LLC); 2021-005588-39 (EudraCT Number)
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Tenofovir; tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Discontinuation of Nucleos(t)ide (NA) Treatment (Experimental): Participants will receive standard of care NA treatment (Entecavir [ETV], Tenofovir Disoproxil Fumarate [TDF], Tenofovir Alafenamide [TAF]) in screening phase (up to 6 weeks) and in baseline visit (Day -1). NA treatment will be discontinued on Day 1 up to 96 weeks (Post-NA discontinuation off-treatment phase). Off-treatment refers to the phase after baseline, in which NA treatment will be discontinued.
  Interventions: Other: Entecavir (ETV); Other: Tenofovir Disoproxil Fumarate (TDF); Other: Tenofovir Alafenamide (TAF)

INTERVENTIONS:
Other: Entecavir (ETV) — ETV will continue throughout screening and will be stopped at baseline.
Other: Tenofovir Disoproxil Fumarate (TDF) — TDF will continue throughout screening and will be stopped at baseline.
Other: Tenofovir Alafenamide (TAF) — TAF will continue throughout screening and will be stopped at baseline.

SUMMARY:
The purpose of this study is to assess the incidence of participants who reach hepatitis B surface antigen (HBsAg) seroclearance after discontinuing nucleos(t)ide analog (NA) therapy in participants with HBsAg less than or equal to (<=) 100 international units per milliliter (IU/mL) and participants with HBsAg greater than (>) 100 IU/mL to <= 500 IU/mL at baseline.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) virus infects the human liver. It consists of a nucleocapsid with hepatitis B core (HBc) protein and a membranous envelope containing hepatitis B surface antigen (HBsAg). Chronic hepatitis B (CHB) virus infection may lead to liver cirrhosis and hepatocellular carcinoma (HCC). Recent guidelines (European Association for the Study of the Liver [EASL] guidelines, Asian Pacific Association for the Study of the Liver [APASL] guidelines) suggest that discontinuation of treatment with nucleos(t)ide analog (NA) (Entecavir [ETV], tenofovir disoproxil fumarate [TDF] or tenofovir alafenamide [TAF]) in non-cirrhotic Hepatitis B e antigen (HBeAg) negative patients after a minimum of three years of viral suppression can trigger changes in virological and immune composition resulting in achieving HBsAg seroclearance (up to 25 percent [%]). The study will be conducted in 3 phases: screening phase (up to 6 weeks), baseline visit (1 day), and post-NA discontinuation phase (up to 96 weeks) which refers to the phase after baseline, in which treatment will be discontinued (off treatment). Discontinuation of NA treatment is considered as study intervention in this study. Collection of core liver biopsy, fine needle aspiration (FNA), and blood samples are considered study investigations/procedures. The participants will be followed for up to 2 years post-NA treatment discontinuation. The total duration of an individual participation will be up to 102 weeks (including up to 6 weeks for screening and baseline).

ELIGIBILITY:
Inclusion Criteria:

* Medically stable on the basis of physical examination, medical history, vital signs, and clinical laboratory tests performed at screening and during the pre-biopsy assessments. If the results of the serum chemistry panel including liver enzymes, blood coagulation, other specific tests, or hematology are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study (in consultation with sponsor)
* Hepatitis B surface antigen (HBsAg) less than or equal to (<=) 500 International units per milliliters (IU/mL) (and greater than [>] 5 IU/mL) at screening
* Hepatitis B e antigen (HBeAg) less than (<) lower limit of quantification and hepatitis B e antibody (HBeAb) positive at screening
* Normal liver ultrasound (at screening or within 3 months before screening [documented evidence])
* Participants must have a body mass index between 18.0 and 35.0 Kilograms per meter square (kg/m^2), extremes included

Exclusion Criteria:

* History of or signs of cirrhosis or portal hypertension (absence of nodules, no smooth liver contour, no normal portal vein, spleen size greater than or equal to [>=] 12 centimeters [cm]) or signs of hepatocellular carcinoma (HCC) or clinically relevant renal abnormalities on an abdominal ultrasound performed within 3 months prior to screening (based on documented evidence, if available) or at the time of screening. In case of suspicious findings on conventional ultrasound the participant may still be eligible if HCC or clinically relevant renal abnormalities have been ruled out by a more specific imaging procedure (contrast enhanced ultrasound, computed tomography [CT] or magnetic resonance imaging [MRI])
* Participant's refusal to accept blood transfusions
* Participants with clinically relevant drug or alcohol abuse within 12 months before screening
* Received an investigational intervention or used an invasive investigational medical device within 3 months before the planned enrollment or is currently enrolled in an investigational study
* Participants of Asian descent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-31 (Estimated); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Hepatitis B Surface Antigen (HBsAg) Seroclearance After Discontinuation of Nucleos(t)ide Analog (NA) Treatment | At Week 24
  Percentage of participants with HBsAg seroclearance after discontinuation of NA treatment will be reported.
Percentage of Participants with HBsAg Seroclearance After Discontinuation of NA Treatment | At Week 48
  Percentage of participants with HBsAg seroclearance after discontinuation of NA treatment will be reported.
Percentage of Participants with HBsAg Seroclearance After Discontinuation of NA Treatment | At Week 96
  Percentage of participants with HBsAg seroclearance after discontinuation of NA treatment will be reported.

SECONDARY OUTCOMES:
Percentage of Participants with Flares | At Week 24, Week 48, and Week 96
  Percentage of participants with flares (virologic, biochemical, and clinical) measured by blood markers (such as HBsAg, hepatitis B virus deoxyribonucleic acid [HBV DNA], and alanine aminotransferase [ALT]) will be reported.
Change from Baseline Over Time in HBsAg Level | Baseline up to 96 weeks
  Change from baseline over time in HBsAg level will be reported.
Change from Baseline Over Time in HBV DNA level | Baseline up to 96 weeks
  Change from baseline over time in HBV DNA level will be reported.
Time to Achieve First HBsAg Seroclearance | Up to 96 weeks
  Time to achieve first HBsAg seroclearance will be reported.
Percentage of Sustained Clinical Responders | At Week 24, Week 48, and Week 96
  Percentage of sustained clinical responders (those with HBsAg seroclearance) will be reported.
Percentage of Participants with HBsAg Seroconversion | At Week 24, Week 48, and Week 96
  Percentage of participants with HBsAg seroconversion will be reported.
Percentage of Participants with Serious Adverse Events (SAEs) | Up to 96 weeks
  SAE is any untoward medical occurrence that results in any of the following conditions that is death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization or results in persistent or significant disability/incapacity.
Percentage of Participants with Abnormalities in Clinical Laboratory Parameters | Up to 96 weeks
  Percentage of participants with abnormalities in clinical laboratory parameters will be reported.
Percentage of Participants Who Meet the NA Re-Treatment Criteria | Up to 96 weeks
  Percentage of participants who meet the NA re-treatment criteria will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency